CLINICAL TRIAL: NCT05996731
Title: Developing a Pipeline to Employ RNA-Seq as a Complementary Diagnostic Tool in Rare Diseases
Acronym: ANTHEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ANTHEM-RNA-Seq
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Atypical Hemolytic Uremic Syndrome; Membranoproliferative Glomerulonephritis; Autosomal Dominant Polycystic Kidney; Healthy
Keywords: Undiagnosed genetic rare diseases; Whole-exome sequencing; RNA-Sequencing; Molecular diagnosis; Skin-derived fibroblasts
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome; Glomerulonephritis, Membranoproliferative; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy subjects (Active Comparator): Five healthy donors will be asked to participate in the study to set up the condition for isolation and culture of skin-derived fibroblasts and to establish the RNA-Seq conditions and profile.
  Interventions: Procedure: Skin biopsy
- Validation cohort (Experimental): To develop a diagnostic pipeline for isolation and sequencing of mRNA from cultured skin fibroblasts, 10 adult patients with known genetic defects affecting RNA levels and/or splicing will be enrolled, as positive controls.
  Interventions: Procedure: Skin biopsy
- Discovery cohort (Experimental): The second group, the discovery cohort, will be composed of 30 undiagnosed symptomatic patients with clinical suspicion of a genetic disease (both children and adults with onset in infancy or early adulthood) referred to the Clinical Research Center for Rare Diseases "Aldo e Cele Daccò", and for which WES analyses did not reveal any causative genetic alteration. To this end, the investigators plan to recruit around 60 patients, their available parents and/or their available informative relatives who will undergo WES, if not previously done. On the basis of literature and their experience, the investigators expect that WES will be resolutive in 40-50% of cases. Consequently, investigators hypothesize to identify 30 patients with a negative WES who will enter the discovery RNA-Seq cohort.
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — A punch biopsy is a 15-minute low-risk procedure performed through a sterile circular blade (usually 3-4 mm) under local anesthesia. Briefly, the instrument is rotated down through the forearm epidermis and dermis perpendicular to its physiological lines of relaxation and into the subcutaneous fat, by producing a cylindrical core. Punch biopsy site can be closed with a single suture and generally produce only a minimal scar.

SUMMARY:
This project aims to identify, through RNA-Seq technology, the genetic alterations underlying undiagnosed rare diseases in pediatric and adult patients with early onset and with negative WES.

* Objective 1: Set up and validate techniques. Set-up and validation of the transcriptome analysis protocol in healthy subjects and in patients with known splicing alterations and/or altered RNA expression.
* Objective 2: Diagnostic phase. Study of splicing alterations and RNA levels in cultured fibroblasts obtained from skin biopsies of patients with rare genetic diseases and negative exome.

Exploratory goals

* Compare the RNA expression profile obtained from skin biopsy-derived fibroblasts with the RNA expression profile from blood. The most relevant results will be validated in qRT-PCR.
* To analyze the transcriptional and protein profile heterogeneity in skin-derived fibroblasts in enrolled subjects.

To explore the effects of genetic (from WES) and transcriptional (from RNA-seq) alterations in participants' plasma and serum.

Healthy controls Five healthy subjects will be recruited from the staff of the Mario Negri Institute for Pharmacological Research. The coded samples will be used to set up the method of isolation and culture of skin fibroblasts and RNA-Seq.

Validation group For the set-up and validation of the skin fibroblast isolation and RNA-Seq procedure, ten adult patients with known diagnosis and with alterations in RNA levels and/or splicing will be recruited as positive controls.

Patients who meet the requirements described above will be contacted by the doctors of the Daccò Center for an interview explaining the project. Those who agree to participate in the study will be asked to sign the informed consent before proceeding with the experimental part.

"Discovery/Exploration" group The exploration cohort will be composed of 30 symptomatic undiagnosed patients with suspected genetic disease (children and adults with infantile onset) belonging to the Clinical Center of the Mario Negri Institute for Pharmacological Research and for whom WES investigations did not reveal causative genetic alterations.

DETAILED DESCRIPTION:
Rare genetic diseases are a very heterogeneous group of diseases, often undiagnosed, for which patients receive only symptomatic treatment. The development of next-generation massive sequencing technology (Next-Generation-Sequencing; NGS) has made it possible to identify many of the genes responsible for these pathologies, allowing the pathogenic mechanisms to be outlined. The most commonly used methods, such as exome sequencing (Whole-Exome Sequencing; WES) or genome sequencing (Whole-Genome Sequencing; WGS), are based on DNA sequencing and allow to identify pathogenic mutations that cause loss of protein functionality, such as stop mutations, large insertions and deletions and the loss of canonical splicing sites. Conversely, the attribution of pathogenicity to an amino acid substitution variant (missense) or a synonymous variant is often questionable and, consequently, such variants are often categorized as Variants of Unknown Significance (VUS). Furthermore, exome sequencing is unable to identify possible pathogenic variants located in non-coding regions, such as non-canonical splice sites or deep intronic variants.

WGS sequencing, while allowing the identification of variants present in the non-coding regions of a gene, is very expensive and produces an enormous amount of data with low pathogenic information. Algorithms to analyze the possible pathogenicity of intronic variants have little predictive power and the pathogenicity of the identified variants must be validated by lengthy and complex functional analyses. Due to these limitations, approximately 50% of patients with rare genetic diseases remain undiagnosed and cannot benefit from the benefits of personalized medicine. Transcriptome sequencing (RNA-Seq) allows to determine variations in the sequence and levels of RNA, providing complementary information to that obtained with WES and WGS, thus improving the efficiency of genetic diagnosis. Splicing alterations, which are among the main causes of genetic diseases and can reside both in deep intronic regions and in coding regions, can be identified through RNA sequencing. Variants in the regulatory regions of the gene, which are able to influence RNA expression levels, can also be highlighted by RNA-Seq. Since RNA expression, in terms of levels and isoforms produced by alternative splicing, is tissue-specific, the most transcriptionally informative biological material is certainly the affected tissue. However, this is not always easy to achieve and the collection can be too invasive for the patient. In these cases it is possible to resort to the use of alternative tissues, such as whole blood or skin biopsies, which have low invasiveness and a broad RNA expression profile. Fibroblasts obtained from skin biopsies, in particular, have proven to be the most reliable, homogeneous and informative alternative matrix for RNA-Seq analysis, in a wide range of pathologies. It has been previously demonstrated that the information obtained from RNA-Seq from skin fibroblasts was superior to that obtained from blood. Furthermore, the analysis of the transcriptome of skin fibroblasts allowed to identify altered levels of transcripts and splicing abnormalities in neuromuscular and neurodevelopmental diseases. This confirmed the efficacy of the use of skin fibroblasts in the diagnosis of genetic pathologies in WES and WGS negative patients. Last but not least, skin fibroblasts can be reprogrammed into other cell types for possible future analyzes.

This project aims to identify, through RNA-Seq technology, the genetic alterations underlying undiagnosed rare diseases in pediatric and adult patients with early onset and with negative WES.

Although NGS is essential for the diagnosis of genetic diseases, its success rates range from 30% to 50%. The advent of RNA-Seq increased the chance of diagnosing genetic diseases from 8% to 36%. Through this project the investigators intend to apply the RNA-Seq method, as an integration of the WES analysis, for the diagnosis of rare genetic diseases:

* Objective 1: Set up and validate techniques. Set-up and validation of the transcriptome analysis protocol in healthy subjects and in patients with known splicing alterations and/or altered RNA expression.
* Objective 2: Diagnostic phase. Study of splicing alterations and RNA levels in cultured fibroblasts obtained from skin biopsies of patients with rare genetic diseases and negative exome.

Exploratory goals.

* To compare the RNA expression profile obtained from skin biopsy-derived fibroblasts with the RNA expression profile from blood. The most relevant results will be validated in qRT-PCR.
* To analyze the transcriptional and protein profile heterogeneity in skin-derived fibroblasts in enrolled subjects.

To explore the effects of genetic (from WES) and transcriptional (from RNA-seq) alterations in participants' plasma and serum.

Healthy controls. Five healthy subjects will be recruited from the staff of the Mario Negri Institute for Pharmacological Research. To ensure the protection of the category of healthy volunteers, it has been envisaged that the enrollment is entrusted to the health personnel of the Daccò Center, who will inform, via email, all the staff of the Institute of the possibility of spontaneously joining the study. No manager or tutor will be involved in the recruitment of volunteers. As a further guarantee of confidentiality, for the purposes of the study, the samples of healthy volunteers will be treated in coded form The coded samples will be used to set up the method of isolation and culture of skin fibroblasts and RNA-Seq.

Validation group. For the set-up and validation of the skin fibroblast isolation and RNA-Seq procedure, ten adult patients with known diagnosis and with alterations in RNA levels and/or splicing will be recruited as positive controls.

Among these, patients affected by atypical Hemolytic-Uremic Syndrome (aHUS), Membranoproliferative Glomerulonephritis (MPGN), Autosomal Dominant Polycystic Kidney (ADPKD) or other rare pathologies previously diagnosed at the Daccò Center will be included, who have given their consent the collection and conservation (UNI EN ISO 9001 since 2016; certification n° 6121) of the samples in the certified biobank (Mario Negri Biological Resources Center - Rare and Kidney Diseases Biobank). Patients who meet the requirements described above will be contacted by the doctors of the Daccò Center for an interview explaining the project. Those who agree to participate in the study will be asked to sign the informed consent before proceeding with the experimental part.

"Discovery/Exploration" group. The exploration cohort will be composed of 30 symptomatic undiagnosed patients with suspected genetic disease (children and adults with infantile onset) belonging to the Clinical Center of the Mario Negri Institute for Pharmacological Research and for whom WES investigations did not reveal causative genetic alterations. To this end the investigators plan to recruit about 60 patients, their parents and more informative family members, if available, who will be analyzed, if not done previously, by WES. Based on the literature and the investigators' experience, it is expected that WES analysis will be curative in 40-50% of cases. Therefore investigators assume to identify 30 patients with negative WES and who will therefore be able to enter the "Discovery/Exploration" cohort.

After signing the informed consent to the collection and storage of samples (UNI EN ISO 9001 since 2016; certification n° 6121) in the certified biobank i.e., the Mario Negri Biological Resources Center - Rare and Renal Diseases Biobank, and after the collection of clinical information, patients will be enrolled in the project.

Blood and skin biopsy samples for DNA and fibroblast isolation will be collected as described below.

For the WES analyses, 3 tubes of 3 ml of whole blood in EDTA will be taken from adults and 2 tubes of 3 ml of whole blood in EDTA from children and stored at -20°C until use. Blood collection will be done at the Mario Negri Institute-Daccò Center.

The WES analyzes will be performed at the Clinical Research Center for Rare Diseases "Aldo e Cele Daccò" or in a specialized external laboratory, selected under our responsibility.

An additional 3 mL aliquot of whole blood will be drawn into TempusTM Blood RNA tubes, for exploratory analysis.

A research biobank containing biological material in the form of blood, serum and plasma will be set up at the "Mario Negri Biological Resource Center - Rare Diseases and Kidney Diseases Biobank".

At the first visit, patients will sign a study-specific consent form, containing specific information and choices regarding participation in the research biobank, including the ability to use the samples in the future for additional research studies.

If subjects give their consent, aliquots of serum and plasma (1 x 2 ml of plasma, 1 x 2 ml of serum) will be collected and stored in coded form in the biobank.

ELIGIBILITY:
Healthy subjects.

Inclusion Criteria:

* Male and female adults
* Written informed consent

Exclusion Criteria:

* Inability to understand the potential risk and benefits of the study
* Legal incapacity

Validation cohort.

Inclusion criteria:

* Male and female adults
* Genetic diseases affecting RNA levels (frameshifts, stop, large deletions, alteration of canonical splicing sites)
* Written informed consent

Exclusion criteria:

* Underage patients
* Inability to understand the potential risk and benefits of the study
* Legal incapacity

Discovery cohort.

Inclusion criteria:

* Male and female patients (children and adults with onset in infancy or early adulthood) with rare genetic undiagnosed diseases
* Patients with no strong candidates based on previous genetic analysis such as WES, but with clinically suspicion of a genetic rare disease
* Written informed consent

Exclusion criteria:

* Inability to understand the potential risk and benefits of the study
* Legal incapacity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Set up and validate the transcriptome analysis procedure in healthy controls and in patients diagnosed with known genetic diseases and with known splice/expression altering variants | At day 0
  WES analyses for DNA isolation
Analyse alterations of mRNA levels and splicing in cultured fibroblasts derived from patients with rare diseases and an inconclusive WES. To investigate the heterogeneity of the transcriptomic and proteomic profile | At day 0
  Skin-derived fibroblasts

CONTACTS AND LOCATIONS:
Overall Officials: Marina Noris, PhD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Centro di Ricerche Cliniche per le Malattie Rare "Aldo e Cele Daccò", Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kremer LS, Bader DM, Mertes C, Kopajtich R, Pichler G, Iuso A, Haack TB, Graf E, Schwarzmayr T, Terrile C, Konarikova E, Repp B, Kastenmuller G, Adamski J, Lichtner P, Leonhardt C, Funalot B, Donati A, Tiranti V, Lombes A, Jardel C, Glaser D, Taylor RW, Ghezzi D, Mayr JA, Rotig A, Freisinger P, Distelmaier F, Strom TM, Meitinger T, Gagneur J, Prokisch H. Genetic diagnosis of Mendelian disorders via RNA sequencing. Nat Commun. 2017 Jun 12;8:15824. doi: 10.1038/ncomms15824. PMID 28604674
- [Background] Lee H, Huang AY, Wang LK, Yoon AJ, Renteria G, Eskin A, Signer RH, Dorrani N, Nieves-Rodriguez S, Wan J, Douine ED, Woods JD, Dell'Angelica EC, Fogel BL, Martin MG, Butte MJ, Parker NH, Wang RT, Shieh PB, Wong DA, Gallant N, Singh KE, Tavyev Asher YJ, Sinsheimer JS, Krakow D, Loo SK, Allard P, Papp JC; Undiagnosed Diseases Network; Palmer CGS, Martinez-Agosto JA, Nelson SF. Diagnostic utility of transcriptome sequencing for rare Mendelian diseases. Genet Med. 2020 Mar;22(3):490-499. doi: 10.1038/s41436-019-0672-1. Epub 2019 Oct 14. PMID 31607746
- [Background] Yepez VA, Mertes C, Muller MF, Klaproth-Andrade D, Wachutka L, Fresard L, Gusic M, Scheller IF, Goldberg PF, Prokisch H, Gagneur J. Detection of aberrant gene expression events in RNA sequencing data. Nat Protoc. 2021 Feb;16(2):1276-1296. doi: 10.1038/s41596-020-00462-5. Epub 2021 Jan 18. PMID 33462443